CLINICAL TRIAL: NCT04574401
Title: A Phase 1 Safety and Efficacy Study of IS-002 Injection in Patients Undergoing Robotic Prostatectomy Using the da Vinci® Surgical System With Firefly® Fluorescent Imaging
Brief Title: A Phase 1 Study of IS-002 Injection in Patients Undergoing Robotic Prostatectomy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: ISI-142325-1
Record Dates: First submitted 2020-09-15; First posted 2020-10-05 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dose escalation (Experimental): Dose-cohort escalation of a single intravenous injection of IS-002 at four different dose levels
  Interventions: Drug: IS-002

INTERVENTIONS:
Drug: IS-002 — Intravenous injection of IS-002 Investigational Drug

SUMMARY:
This is a Phase 1, single-site, interventional clinical trial evaluating the safety and efficacy of IS-002 intravenous (IV) injection for fluorescent identification and delineation of the positive cancer margins and metastatic lymph nodes during prostatectomy surgery using the da Vinci® X/Xi Surgical System with Firefly® Fluorescent Imaging.

ELIGIBILITY:
Inclusion Criteria:

* Subject is between the ages of 18 and 75.
* Subject has a confirmed adenocarcinoma by histology of the prostate.
* Subject has CAPRA > 6, or T3 a or b disease on imaging (TRUS and/or MRI), or regional lymphadenopathy suspicious for nodal metastases
* Subject is scheduled to undergo robotic prostatectomy with extended pelvic lymph node dissection (ePLND) using an da Vinci® X/Xi Surgical System with Firefly® Fluorescent Imaging.
* Subject is willing and able to provide informed consent
* Subject is considered capable of complying with study procedures and of understanding a written informed consent document.
* Subject must be treatment naïve (not having received neo-adjuvant therapy, radiation therapy, hormonal therapy, androgen deprivation therapy within the last 4 months excluding Finasteride, Dutasteride, or other 5 alpha reductase inhibitors, or focal ablation techniques)

Exclusion Criteria:

* Subject has known active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection
* Subject is currently participating in and receiving study therapy or has participated in a study of an investigational agent within the past 6 months; is receiving study therapy or is involved in a significant risk investigational device study within the past 6 months
* Subject has any other condition or personal circumstance that, in the judgment of the Investigator, might interfere with the collection of complete quality data or represents an unacceptable safety profile
* Subject has a known history of bone metastasis documented on the basis of bone scans and/or biopsy
* Subject has a known history of acute or chronic liver or kidney disease

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 24 (Actual)
Dates: Start 2020-10-10 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2021-09-20 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events as assessed by CTCAE v5.0 | 14 days
  Number of participants treated with IS-002 with treatment-emergent adverse events as assessed by CTCAE v5.0

SECONDARY OUTCOMES:
IS-002 Maximum Plasma Concentration (Cmax) | -5 minutes (pre-study drug), 5 minutes, 15 minutes, 30 minutes, 60 minutes, 2 hours, 4 hours, 6 hours, 24 hours
  Maximum Plasma Concentration (Cmax) of IS-002
IS-002 Half-Life (t½) | -5 minutes (pre-study drug), 5 minutes, 15 minutes, 30 minutes, 60 minutes, 2 hours, 4 hours, 6 hours, 24 hours
  Half-Life (t½) of IS-002
IS-002 Clearance (CL) | -5 minutes (pre-study drug), 5 minutes, 15 minutes, 30 minutes, 60 minutes, 2 hours, 4 hours, 6 hours, 24 hours
  Clearance (CL) of IS-002
IS-002 Area Under the Plasma Concentration Versus Time Curve (AUC) | -5 minutes (pre-study drug), 5 minutes, 15 minutes, 30 minutes, 60 minutes, 2 hours, 4 hours, 6 hours, 24 hours
  Area Under the Plasma Concentration Versus Time Curve (AUC) of IS-002

OTHER OUTCOMES:
The number of subjects with above-background IS-002 fluorescent signal observed on the prostate surface that is confirmed as a positive surgical margin through pathological confirmation of malignant tissue via hematoxylin and eosin stain. | 30 days
  An exploratory outcome measure of cancer fluorescent signal levels relative to normal tissue (tumor-to-background ratios) confirmed with gold standard histopathology
The number of lymph nodes with IS-002 fluorescent signal that contain metastatic disease as confirmed through pathological confirmation of malignant tissue via hematoxylin and eosin stain. | 30 days
  An exploratory outcome measure of cancer fluorescent signal levels relative to normal tissue (tumor-to-background ratios) confirmed with gold standard histopathology

CONTACTS AND LOCATIONS:
Locations (1):
- UCSF Medical Center, Mission Bay, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No